CLINICAL TRIAL: NCT00818532
Title: Corneal Astigmatism Measurement Study
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: P-08-04
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2009-07

CONDITIONS: Astigmatism
Keywords: Corneal astigmatism; Low diopter; Corneal measurement; Corneal astigmatism < 1 Diopter
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Measurement device

SUMMARY:
To assess which commercially available measurement device is most accurate in measuring low (< 1.0 D) degrees of corneal astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age and older
* Proof of eye exam within the last 3 months
* Corneal astigmatism of <1.0 diopter

Exclusion Criteria:

* Prior history of refractive or corneal surgery
* Corneal trauma/disease
* Intraocular surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Measurement of corneal power | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States